CLINICAL TRIAL: NCT06626061
Title: Promotion of Mental Health and Prevention of Burnout Among Caregivers at CHU Grenoble Alpes (CHUGA) and CH Métropole Savoie (CHMS) Through a Stress Management Intervention Based on Cognitive Behavioral Therapies.
Brief Title: Evaluation of the CBSM Program Online and in Person to Reduce Caregiver Burnout
Acronym: Caregiver-CBSM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 38RC24.0301; 2024-A01832-45 (Other: ID RCB)
Record Dates: First submitted 2024-09-26; First posted 2024-10-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Burnout, Caregiver
Keywords: Mental health promotion; Caregiver Burnout; CBT Intervention; Stress Management
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CBSM Intervention in In-Person Group Format (Experimental): * 8 CBSM sessions
  * The sessions will take place in a group setting, face-to-face, within the institution.
  Interventions: Behavioral: Cognitive Behavioral Stress management in in person group Format
- Hybrid CBSM Intervention (Experimental): * 8 CBSM sessions
  * This format combines podcasts to listen to, along with three online sessions via video conferencing (at the beginning, middle, and end of the program).
  Interventions: Behavioral: Cognitive Behavioral Stress management Hybrid Format
- Delayed CBSM Intervention (No Intervention): Participants will participate in the program at a delayed time to form a control group.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress management in in person group Format — The CBSM sessions will be delivered to participants in groups of ten, totaling eight sessions, each focused on a specific theme related to stress management. All participants will attend the complete sessions in person.
  Arms: CBSM Intervention in In-Person Group Format
Behavioral: Cognitive Behavioral Stress management Hybrid Format — The CBSM (hybrid) sessions will be offered to participants online, including a total of eight video modules, each dedicated to a specific theme related to stress management. Participants will also have access to three interactive virtual sessions, summary sheets in PDF format, and audio recordings for relaxation.
  Arms: Hybrid CBSM Intervention

SUMMARY:
Professional burnout is a common syndrome among healthcare workers, impacting both their well-being and the quality of care provided . It is characterized by emotional exhaustion, depersonalization, and a reduced sense of personal accomplishment.

This multicenter study evaluates the effectiveness of the Cognitive Behavioral Stress Management (CBSM) program in preventing burnout. This intervention, based on cognitive-behavioral techniques, integrates stress management tools and relaxation exercises over eight 2-hour sessions. The study aims to recruit 200 healthcare workers, divided into three groups: in-person intervention, hybrid format (videos + videoconferences), and delayed intervention (in-person/hybrid), across two hospital centers (CHUGA and CHMS). Data will be collected at three time points (M0, M3, M6), with emotional exhaustion (MBI) as the primary outcome, supplemented by measures of individual, relational, and organizational factors.

By comparing different intervention modalities (in-person vs. hybrid, immediate vs. delayed), this research will provide practical recommendations to enhance burnout prevention strategies in the hospital setting.

DETAILED DESCRIPTION:
This project aims to evaluate the effectiveness of the Cognitive Behavioral Stress Management (CBSM) program in preventing burnout, a widespread issue among healthcare professionals. Burnout, particularly characterized by emotional exhaustion, depersonalization, and reduced personal accomplishment, has severe consequences on caregivers' mental and physical health as well as the quality of care provided. In this context, the CBSM program, originally developed for patients, has been modified and adapted specifically to meet the needs of healthcare professionals. It is a multidimensional program combining various techniques such as relaxation, cognitive and emotional management, coping strategies and enhancement of social support and assertiveness. Numerous previous studies have demonstrated the effectiveness of CBSM in reducing stress, anxiety, and depressive symptoms, as well as in improving the long-term quality of life of participants.

The current project plans to form 12 groups of 10 people, split between the two institutions, with two intervention modalities: in-person group sessions and a hybrid format. The latter includes podcasts and three virtual sessions (at the beginning, middle, and end of the program). Participants, whether medical or non-medical staff, will complete standardized questionnaires before the intervention begins (M0), at the end of the intervention (M3), and six months later (M6). Data collection will take place from May 2025 to December 2026, with the last inclusion scheduled for October 2026.

All data will be collected via questionnaires:

* The Maslach Burnout Inventory (MBI), which will assess the three dimensions of burnout: emotional exhaustion, depersonalization, and personal accomplishment.
* The Perceived Stress Scale (PSS-14), which will measure the participants' perceived stress levels.
* The Hospital Anxiety and Depression Scale (HADS), which will evaluate symptoms of anxiety and depression among participants.
* The Professional Quality of Life Scale (ProQOL), which will assess participants' professional quality of life.
* The Ruminative Response Scale (RRS), which will evaluate participants' tendencies toward rumination.
* The Coping Flexibility Scale-Revised (CFS-R), which will measure individuals' ability to evaluate the effectiveness of their coping strategies and to replace them when they are not effective.
* A questionnaire on program satisfaction and adherence.
* Sociodemographic data (age, gender, years of experience in the profession) to identify variations in the effectiveness of the intervention based on caregivers' profiles.
* Questions regarding perceptions of working conditions.
* One item measuring sleep quality.
* Two items measuring social support at work and outside of work.

The expected outcomes of this study aim to enrich the scientific literature on burnout prevention and stress management in healthcare professionals, providing recommendations on best practices to be disseminated across healthcare institutions. The results will also be used to develop continuing education programs designed to strengthen healthcare professionals psychosocial skills.

ELIGIBILITY:
Inclusion criteria :

* Be a healthcare professional.
* Be a volunteer.
* Work at CHUGA or CHMS.
* Be available to attend program sessions (in-person or hybrid).

Exclusion criteria:

* Protected persons (articles L1121-5 to L1121-8 of the Public Health Code), except for pregnant women for whom a benefit is expected in relation to a foreseeable minor risk for the pregnant woman or the unborn child.
* Students in health-related fields.
* Individuals with difficulties in understanding the French language.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Score of the Emotional Exhaustion Dimension of the Maslach Burnout Inventory (MBI) | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  The scores for the emotional exhaustion dimension of the Maslach Burnout Inventory (MBI) range from 0 to 54. A higher score indicates a higher level of emotional exhaustion.

SECONDARY OUTCOMES:
Scores of Depersonalization and Personal Accomplishment from the Maslach Burnout Inventory (MBI). | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  The scores for the depersonalization dimension of the Maslach Burnout Inventory (MBI) range from 0 to 30. A higher score indicates a higher level of depersonalization. For the personal accomplishment dimension, scores range from 0 to 48, where a lower score signifies reduced personal accomplishment.
Perceived stress assessed by the Perceived Stress Scale (PSS-14) | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Anxiety and depression assessed by the Hospital Anxiety and Depression Scale (HADS). | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  The Hospital Anxiety and Depression Scale (HADS) assesses two dimensions: anxiety (HADS-A) and depression (HADS-D), each with a minimum score of 0 and a maximum score of 21. Higher score indicates significant clinical symptoms of anxiety or depression.
Rumination assessed by the Rumination Response Scale. (RRS) | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  Individual scores on the RSS can range from 5 to 20 for each subscale. (Brooding and reflexion) Higher score reflects a high tendency to ruminate.
Quality of life at work assessed by the Professional Quality of Life (ProQOL) Scale. | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  Individual scores on the ProQOL can range from 0 to 30. Higher score indicates the following: for Compassion Satisfaction (CS), it reflects a strong joy in helping others; for Burnout (BO), it signifies a high level of professional exhaustion; and for Secondary Traumatic Stress (STS), it denotes a significant level of secondary traumatic stress related to others' experiences.
working conditions questionnaire | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  Individual scores on the working conditions questionnaire can range from 0 to 90. Higher score indicates good working conditions.
socio-demographic data questionnaire | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  Age, gender, type of hospital service...
A questionnaire on program satisfaction and adherence. | Month 3; Month 6 for the immediate intervention group and Month 6; Month 9 for the delayed intervention group
  It will assess participants' level of satisfaction with the program (e.g., content relevance, usefulness, delivery format) and their engagement (e.g., attendance, completion of exercises). This questionnaire will help identify areas for improvement and better understand participants' experience with the intervention.
Coping flexibility | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  12-item self-report measure assessing individuals' ability to evaluate and adjust their coping strategies based on their effectiveness. It reflects the dynamic process of stress management, where a person may modify or abandon a strategy if it proves ineffective or harmful. Participants rate each item on a 4-point scale (0 = not applicable to 3 = very applicable).
  The scale includes three subdimensions:
  Abandonment - ability to discontinue ineffective coping strategies Re-coping - ability to generate and apply alternative strategies Meta-coping - awareness and evaluation of coping effectiveness
  A higher total score indicates greater coping flexibility.
1 item measuring sleep quality. | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  "Over the past month, how would you rate the overall quality of your sleep?" 0 = Very poor to 10 = Very good
2 items measuring social support: | Month 0; Month 3; Month 6 for the immediate intervention group and Month 0; Month 3; Month 6; Month 9 for the delayed intervention group
  "Overall, to what extent do you feel supported outside of work (family, friends, etc.)?"( 0 = Very little support to 10 = Very well supported)
  "Overall, to what extent do you feel supported at work?" ( 0 = Very little support to 10 = Very well supported)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Gauchet, Professor, Study Director — Université Savoie Mont Blanc; Nour Chiboub, doctoral student, Study Director — Université Savoie Mont Blanc; Anne-Sophie Wasmer, Doctor, Study Director — Centre Hospitalier Métropole Savoie (Chambéry); Véronique Bollongeat, Doctor, Study Director — Centre Hospitalier Universitaire Grenoble Alpes; Jean-Luc Bosson, Professor, Study Chair — Centre Hospitalier Universitaire Grenoble Alpes
Locations (2):
- France (2):
  - Centre Hospitalier Métropole Savoie (CHMS), Chambéry, France
  - Centre hospitalier Grenoble Alpes (CHUGA), Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoni MH, Lechner S, Diaz A, Vargas S, Holley H, Phillips K, McGregor B, Carver CS, Blomberg B. Cognitive behavioral stress management effects on psychosocial and physiological adaptation in women undergoing treatment for breast cancer. Brain Behav Immun. 2009 Jul;23(5):580-91. doi: 10.1016/j.bbi.2008.09.005. Epub 2008 Sep 20. PMID 18835434
- [Background] Lopez C, Antoni M, Penedo F, Weiss D, Cruess S, Segotas MC, Helder L, Siegel S, Klimas N, Fletcher MA. A pilot study of cognitive behavioral stress management effects on stress, quality of life, and symptoms in persons with chronic fatigue syndrome. J Psychosom Res. 2011 Apr;70(4):328-34. doi: 10.1016/j.jpsychores.2010.11.010. Epub 2011 Jan 15. PMID 21414452
- [Background] Stagl JM, Antoni MH, Lechner SC, Bouchard LC, Blomberg BB, Gluck S, Derhagopian RP, Carver CS. Randomized controlled trial of cognitive behavioral stress management in breast cancer: a brief report of effects on 5-year depressive symptoms. Health Psychol. 2015 Feb;34(2):176-80. doi: 10.1037/hea0000125. Epub 2014 Jul 28. PMID 25068452
- [Background] Traeger L, Penedo FJ, Benedict C, Dahn JR, Lechner SC, Schneiderman N, Antoni MH. Identifying how and for whom cognitive-behavioral stress management improves emotional well-being among recent prostate cancer survivors. Psychooncology. 2013 Feb;22(2):250-9. doi: 10.1002/pon.2074. Epub 2011 Sep 19. PMID 21932396
- [Background] Antoni MH, Lechner SC, Kazi A, Wimberly SR, Sifre T, Urcuyo KR, Phillips K, Gluck S, Carver CS. How stress management improves quality of life after treatment for breast cancer. J Consult Clin Psychol. 2006 Dec;74(6):1143-52. doi: 10.1037/0022-006X.74.6.1152. PMID 17154743
- [Background] Antoni MH, Wimberly SR, Lechner SC, Kazi A, Sifre T, Urcuyo KR, Phillips K, Smith RG, Petronis VM, Guellati S, Wells KA, Blomberg B, Carver CS. Reduction of cancer-specific thought intrusions and anxiety symptoms with a stress management intervention among women undergoing treatment for breast cancer. Am J Psychiatry. 2006 Oct;163(10):1791-7. doi: 10.1176/ajp.2006.163.10.1791. PMID 17012691
- [Background] Baumgarten C, Michinov E, Rouxel G, Bonneterre V, Gay E, Roche PH. Personal and psychosocial factors of burnout: A survey within the French neurosurgical community. PLoS One. 2020 May 29;15(5):e0233137. doi: 10.1371/journal.pone.0233137. eCollection 2020. PMID 32469930
- [Background] Bocerean C, Dupret E. A validation study of the Hospital Anxiety and Depression Scale (HADS) in a large sample of French employees. BMC Psychiatry. 2014 Dec 16;14:354. doi: 10.1186/s12888-014-0354-0. PMID 25511175
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Dres M, Copin MC, Cariou A, Mathonnet M, Gaillard R, Shanafelt T, Riou B, Darmon M, Azoulay E. Job Strain, Burnout, and Suicidal Ideation in Tenured University Hospital Faculty Staff in France in 2021. JAMA Netw Open. 2023 Mar 1;6(3):e233652. doi: 10.1001/jamanetworkopen.2023.3652. PMID 36976563
- [Background] Fekete EM, Antoni MH, Schneiderman N. Psychosocial and behavioral interventions for chronic medical conditions. Curr Opin Psychiatry. 2007 Mar;20(2):152-7. doi: 10.1097/YCO.0b013e3280147724. PMID 17278914
- [Background] Hammerfald K, Eberle C, Grau M, Kinsperger A, Zimmermann A, Ehlert U, Gaab J. Persistent effects of cognitive-behavioral stress management on cortisol responses to acute stress in healthy subjects--a randomized controlled trial. Psychoneuroendocrinology. 2006 Apr;31(3):333-9. doi: 10.1016/j.psyneuen.2005.08.007. Epub 2005 Sep 23. PMID 16183205
- [Background] Heritage B, Rees CS, Hegney DG. The ProQOL-21: A revised version of the Professional Quality of Life (ProQOL) scale based on Rasch analysis. PLoS One. 2018 Feb 28;13(2):e0193478. doi: 10.1371/journal.pone.0193478. eCollection 2018. PMID 29489875
- [Background] Lefevre H, Stheneur C, Cardin C, Fourcade L, Fourmaux C, Tordjman E, Touati M, Voisard F, Minassian S, Chaste P, Moro MR, Lachal J. The Bulle: Support and Prevention of Psychological Decompensation of Health Care Workers During the Trauma of the COVID-19 Epidemic. J Pain Symptom Manage. 2021 Feb;61(2):416-422. doi: 10.1016/j.jpainsymman.2020.09.023. Epub 2020 Sep 19. PMID 32961219
- [Background] Marine A, Ruotsalainen J, Serra C, Verbeek J. Preventing occupational stress in healthcare workers. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD002892. doi: 10.1002/14651858.CD002892.pub2. PMID 17054155
- [Background] McClafferty H, Brown OW; Section on Integrative Medicine; Committee on Practice And Ambulatory Medicine; Section on Integrative Medicine. Physician health and wellness. Pediatrics. 2014 Oct;134(4):830-5. doi: 10.1542/peds.2014-2278. PMID 25266440
- [Background] Moeini B, Hazavehei SM, Hosseini Z, Aghamolaei T, Moghimbeigi A. The Impact of Cognitive-Behavioral Stress Management Training Program on Job Stress in Hospital Nurses: Applying PRECEDE Model. J Res Health Sci. 2011 Nov 4;11(2):114-20. PMID 22911962
- [Background] Muller L, Spitz E. [Multidimensional assessment of coping: validation of the Brief COPE among French population]. Encephale. 2003 Nov-Dec;29(6):507-18. French. PMID 15029085
- [Background] Pospos S, Young IT, Downs N, Iglewicz A, Depp C, Chen JY, Newton I, Lee K, Light GA, Zisook S. Web-Based Tools and Mobile Applications To Mitigate Burnout, Depression, and Suicidality Among Healthcare Students and Professionals: a Systematic Review. Acad Psychiatry. 2018 Feb;42(1):109-120. doi: 10.1007/s40596-017-0868-0. Epub 2017 Dec 18. PMID 29256033
- [Background] Rainforth MV, Schneider RH, Nidich SI, Gaylord-King C, Salerno JW, Anderson JW. Stress reduction programs in patients with elevated blood pressure: a systematic review and meta-analysis. Curr Hypertens Rep. 2007 Dec;9(6):520-8. doi: 10.1007/s11906-007-0094-3. PMID 18350109
- [Background] Reis RS, Hino AA, Anez CR. Perceived stress scale: reliability and validity study in Brazil. J Health Psychol. 2010 Jan;15(1):107-14. doi: 10.1177/1359105309346343. PMID 20064889
- [Background] Servant D, Rougegrez L, Barasino O, Demarty AL, Duhamel A, Vaiva G. [Interest of computer-based cognitive behavioral stress management. Feasability of the Seren@ctif program]. Encephale. 2016 Oct;42(5):415-420. doi: 10.1016/j.encep.2016.03.010. Epub 2016 Apr 25. French. PMID 27126141
- [Background] Stagl JM, Bouchard LC, Lechner SC, Blomberg BB, Gudenkauf LM, Jutagir DR, Gluck S, Derhagopian RP, Carver CS, Antoni MH. Long-term psychological benefits of cognitive-behavioral stress management for women with breast cancer: 11-year follow-up of a randomized controlled trial. Cancer. 2015 Jun 1;121(11):1873-81. doi: 10.1002/cncr.29076. Epub 2015 Mar 23. PMID 25809235
- [Background] Tatrow K, Montgomery GH. Cognitive behavioral therapy techniques for distress and pain in breast cancer patients: a meta-analysis. J Behav Med. 2006 Feb;29(1):17-27. doi: 10.1007/s10865-005-9036-1. Epub 2006 Jan 7. PMID 16400532
- [Background] Terp U, Bisholt B, Hjarthag F. Not Just Tools to Handle It: A Qualitative Study of Nursing Students' Experiences From Participating in a Cognitive Behavioral Stress Management Intervention. Health Educ Behav. 2019 Dec;46(6):922-929. doi: 10.1177/1090198119865319. Epub 2019 Aug 8. PMID 31394927
- [Background] Vancappel A, Jansen E, Ouhmad N, Desmidt T, Etain B, Bergey C, d'Ussel M, Krebs MO, Paquet C, Reveillere C, Hingray C, El-Hage W. Psychological Impact of Exposure to the COVID-19 Sanitary Crisis on French Healthcare Workers: Risk Factors and Coping Strategies. Front Psychiatry. 2021 Nov 18;12:701127. doi: 10.3389/fpsyt.2021.701127. eCollection 2021. PMID 34867507